CLINICAL TRIAL: NCT00000992
Title: Pilot Study to Determine the Feasibility of Itraconazole for Suppression of Relapse of Disseminated Histoplasmosis in Patients With the Acquired Immunodeficiency Syndrome
Brief Title: A Study of Itraconazole in Preventing the Return of Histoplasmosis, a Fungal Infection, in Patients With AIDS
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Masking: None | Purpose: Treatment
Other Study IDs: ACTG 084; 11059 (Registry Identifier: DAIDS ES Registry Number)
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-11-01 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections; Histoplasmosis
Keywords: AIDS-Related Opportunistic Infections; Ketoconazole; Histoplasmosis; Drug Evaluation; Antifungal Agents; Acquired Immunodeficiency Syndrome
MeSH Terms: conditions — HIV Infections; Histoplasmosis; AIDS-Related Opportunistic Infections; Acquired Immunodeficiency Syndrome | interventions — Itraconazole

INTERVENTIONS:
Drug: Itraconazole

SUMMARY:
To test the effectiveness of itraconazole in preventing the recurrence of disseminated histoplasmosis in AIDS patients.

Histoplasmosis is a serious opportunistic infection in patients with AIDS. Amphotericin B has been used to treat the infection. Although the response to this treatment is generally good, up to 90 percent of AIDS patients who have taken amphotericin B to treat their histoplasmosis infection will have a relapse (that is, they will get the disease again) within 12 months following treatment. Ketoconazole has been used to prevent relapse, but available information suggests that up to 50 percent of AIDS patients relapse even with ketoconazole treatment. A more effective therapy to prevent recurrence is needed. Itraconazole has been used successfully to treat disseminated histoplasmosis in non-AIDS patients and it is hoped that it may be more effective in preventing histoplasmosis relapse.

DETAILED DESCRIPTION:
Histoplasmosis is a serious opportunistic infection in patients with AIDS. Amphotericin B has been used to treat the infection. Although the response to this treatment is generally good, up to 90 percent of AIDS patients who have taken amphotericin B to treat their histoplasmosis infection will have a relapse (that is, they will get the disease again) within 12 months following treatment. Ketoconazole has been used to prevent relapse, but available information suggests that up to 50 percent of AIDS patients relapse even with ketoconazole treatment. A more effective therapy to prevent recurrence is needed. Itraconazole has been used successfully to treat disseminated histoplasmosis in non-AIDS patients and it is hoped that it may be more effective in preventing histoplasmosis relapse.

AIDS patients who have been successfully treated with amphotericin B for an acute first episode of disseminated histoplasmosis are selected for treatment. They receive daily oral doses of itraconazole for a total of 52 weeks. Patients who do not experience significant toxicity related to the drug may continue to receive itraconazole until the last patient completes 52 weeks of itraconazole therapy or has the study drug discontinued prior to completing 52 weeks of therapy. AMENDED: Patients will be treated for a minimum of 52 weeks. Patients who complete the 52 weeks and remain on the study drug will continue to be followed. If itraconazole becomes licensed for histoplasmosis, study drug must be discontinued at the end of 52 weeks of therapy or at the time of licensure for patients who have received more than 52 weeks of therapy.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Itraconazole therapy must begin no more than 6 weeks after discontinuing primary amphotericin B therapy; itraconazole therapy may begin immediately after stopping the primary therapy with amphotericin B.

Allowed:

* Oral contraceptives.
* Methadone.
* Narcotics.
* Acyclovir.
* Acetaminophen.
* Sulfonamides.
* Trimethoprim / sulfamethoxazole.
* Aerosolized pentamidine for Pneumocystis carinii pneumonia (PCP) or PCP prophylaxis (patients with a total CD4+ count < 200 or a history of PCP should receive PCP prophylaxis).
* Treatment IND drugs.
* Zidovudine.
* Topical antifungals.
* Discouraged:
* Antacids.
* Sucralfate.
* H2 blockers.

Concurrent Treatment:

Allowed:

* Radiation therapy for mucocutaneous Kaposi's sarcoma.

Prior Medication:

Required:

* Prior treatment with amphotericin B for disseminated histoplasmosis:
* minimum total dose of 15 mg/kg for patients < 67 kg, or 1 g for patients > 67 kg; must have been administered over 6 months or less.

Allowed:

* Amphotericin B as maintenance therapy for a maximum of 6 weeks following completion of primary therapy.
* Zidovudine.
* Prophylaxis for Pneumocystis carinii pneumonia.

Exclusion Criteria

Co-existing Condition:

Patients with the following conditions are excluded:

* History of allergy to, or intolerance of, imidazoles or azoles.
* Clinical findings of active histoplasmosis.
* Histoplasmosis of the central nervous system.
* Inability to take oral medications reliably or severe malabsorption syndrome.
* Malignancies requiring cytotoxic therapy.
* Culture-proven systemic Mycobacterium tuberculosis, Mycobacterium avium-intracellulare, coccidioidomycosis, or cryptococcosis.

Concurrent Medication:

Excluded:

* Amphotericin B as maintenance therapy.
* Immunostimulants.
* Ketoconazole.
* Systemic antifungals.
* Steroids in excess of physiologic replacement doses.
* Cytotoxic chemotherapy.
* Investigational agents not specifically allowed.
* Antacids for 4 hours before and 4 hours after itraconazole.

Concurrent Treatment:

Excluded:

* Lymphocyte replacement.

Patients with the following conditions are excluded:

* History of allergy to, or intolerance of, imidazoles or azoles.
* Clinical findings of active histoplasmosis.
* Histoplasmosis of the central nervous system.
* Inability to take oral medications reliably or severe malabsorption syndrome.
* Malignancies requiring cytotoxic therapy.
* Culture-proven systemic Mycobacterium tuberculosis, Mycobacterium avium-intracellulare, coccidioidomycosis, or cryptococcosis.

Prior Medication:

Excluded within 30 days of study entry:

* Immunostimulants.
* Ketoconazole.
* Systemic antifungals.
* Steroids in excess of physiologic replacement doses.
* Cytotoxic chemotherapy.

Prior Treatment:

Excluded:

* Lymphocyte replacement.

Risk Behavior:

Excluded:

* Patients who in the opinion of the investigator would be undependable with regard to adherence to protocol.

Inclusion criteria are:

* HIV infection documented by presence of antibody, by ELISA with Western blot confirmation, or serum p24 antigen, or by recovery of HIV in culture.
* Acute first episode of disseminated histoplasmosis documented by recovery and identification of H. capsulatum from cultures obtained from extrapulmonary sites.
* Oriented to person, place, and time, and able to give written informed consent.

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30
Dates: Study Completion 1992-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: LJ Wheat, Study Chair
Locations (8):
- United States (8):
  - USC CRS, Los Angeles, California
  - Northwestern University CRS, Chicago, Illinois
  - Indiana Univ. School of Medicine, Infectious Disease Research Clinic, Indianapolis, Indiana
  - Tulane Med. Ctr. - Charity Hosp. of New Orleans, ACTU, New Orleans, Louisiana
  - Washington U CRS, St Louis, Missouri
  - Cornell University A2201, New York, New York
  - Univ. of Cincinnati CRS, Cincinnati, Ohio
  - Pitt CRS, Pittsburgh, Pennsylvania

REFERENCES:
- [Background] Wheat J, Hafner R, Wulfsohn M, Spencer P, Squires K, Powderly W, Wong B, Rinaldi M, Saag M, Hamill R, Murphy R, Connolly-Stringfield P, Briggs N, Owens S; National Institute of Allergy and Infectious Diseases Clinical Trials and Mycoses Study Group Collaborators. Prevention of relapse of histoplasmosis with itraconazole in patients with the acquired immunodeficiency syndrome. Ann Intern Med. 1993 Apr 15;118(8):610-6. doi: 10.7326/0003-4819-118-8-199304150-00006. PMID 8383934